CLINICAL TRIAL: NCT04506944
Title: The Epidemiology Of Scrub Typhus And Rickettsial Infections In A Highly Endemic Rural Setting In South India: Population-Based Cohort Study
Brief Title: The Epidemiology of Rickettsial Infections in South India: Cohort Study
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Medical Research Council (Other Government); Christian Medical College, Vellore, India (Other); Mahidol Oxford Tropical Medicine Research Unit (Other); Australian Rickettsial Reference Laboratory (Unknown)
Responsible Party: Sponsor
Other Study IDs: MRC typhus cohort 1
Record Dates: First submitted 2020-08-07; First posted 2020-08-10 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Scrub Typhus; Spotted Fever; India; Murine Typhus
MeSH Terms: conditions — Scrub Typhus; Spotted Fever Group Rickettsiosis; Typhus, Endemic Flea-Borne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples from human participants: serum for serological testing, buffy coat for rickettsia PCR Eschar and skin biopsies for rickettsia PCR
  Arthropod vector samples: PCR for rickettsia Rodent tissue samples: PCR for rickettsia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- General population: Whole population of scrub typhus endemic villages
  Interventions: Other: No intervention
- hospital case population: cases recruited at study clinics who are not enrolled in general population cohort
  Interventions: Other: No intervention
- Serological cohort: random subset of 4000 participants above the age of 10 drawn from general population cohort
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No specific exposure is explored.

SUMMARY:
There is enough evidence to suggest that scrub typhus and spotted fever group rickettsioses are common causes of febrile illness in India. Serological evidence also exists for murine typhus, but is rarely tested for. Incidence, risk factors, clinical features and molecular epidemiology of these three infections are poorly understood. Delays in disease recognition and treatment may cause thousands of preventable deaths across India.

The objectives of the research are to determine the incidence and risk factors of scrub typhus, spotted fever and murine typhus by severity, to determine clinical features of these neglected and often unrecognized infections. Further to study the effect of previous infection on incidence and severity of subsequent infections. Finally to study the association between vector parameters and scrub typhus risk.

Enrolled will be 30,000 individuals who will be followed up for the development of fever using active and passive surveillance. Active surveillance will include household screening every 3-6 weeks. Fever cases occuring in the past two months will be tested for Scrub typhus, murine typhus and spotted fever IgG/IgM. 4000 individuals will be followed up by annual serological testing to identify asymptomatic infections. Participants notifying the study team with ongoing fever will undergo blood testing for acute diagnosis of rickettsial infection (IgM, PCR). In addition, we will enroll fever cases at study clinics who are not part of the main cohort. The research includes spatial and socio-economic risk factor analysis. Rodents carrying mite larvae will be trapped to compare the intensity of mite infestation between areas of high and low risk for human scrub typhus.

The data on incidence, burden of disease and environmental determinants of scrub typhus, spotted fever and murine typhus will be used for health care planning and information campaigns for the public and medical professionals.

DETAILED DESCRIPTION:
The aim of the cohort study is to better understand the epidemiology, sero-epidemiology and transmission of scrub typhus, murine typhus and tick-borne spotted fever. The overall focus of the work will be on scrub typhus, being the most important of the three from the public health perspective. We aim to determine the "severity pyramid" of serological, symptomatic and severe infection. The results from this study will help clinicians to understand the natural course of scrub typhus infection, health policy makers to estimate the global burden and the scope for community-based interventions, and immunologists to better understand the immunogenicity of single and repeat infections.

The specific objectives are to:

1. Estimate the incidence of symptomatic and severe scrub typhus infection in the community.
2. Estimate the incidence of serological (asymptomatic) scrub typhus infection.
3. Estimate the effect of previous scrub typhus infection (sero-positive at baseline) on the risk of subsequent infection and disease severity (subclinical vs clinically apparent). This includes the effect of antibodies in mothers on the risk of severe infection in young children via residual maternal antibodies.
4. Estimate the effect of potential risk factors such as age, gender, occupation, water/sanitation access and comorbidity on the risk of scrub typhus infection.
5. Estimate the effect of spatial-temporal risk factors for scrub typhus by identifying high risk areas, accounting for human population density and land use.
6. Compare the rate of rodent trappings and vector parameters of chiggers between high risk and low risk areas identified under 5).
7. Estimate the disease burden associated with scrub typhus and the economic impact of scrub typhus in terms of loss of earnings and health expenditure.
8. Estimate the incidence of asymptomatic and symptomatic murine typhus and spotted fever infection and explore associated socio-demographic, spatial and vector-related risk factors.

STUDY OVERVIEW

The study will be a population-based cohort study over two years (i.e. two scrub typhus seasons) in about 30,000 people living in approximately 40 villages with a sero-prevalence of at least 15% (see flow diagram above). These individuals will be followed-up through active surveillance for recent febrile illnesses (clinical cohort). For passive surveillance, participants will be encouraged to notify the study team in case of fever or come to one of 4 local study clinics. At study clinics we will also enrol fever cases who are not part of the clinical cohort, i.e. have not been enrolled prior to their fever. The study will include a smaller cohort (sero-cohort) for serological surveillance of 4000 people drawn from the 30,000 people of the clinical cohort. Longitudinal serological surveys linked to active surveillance are essential to estimate true attack rates unbiased by disease severity. The sero-cohort will consist of three annual blood testing in the same group of participants over two scrub typhus seasons (baseline, inter-season, endline).

Target population- A pilot study showed that scrub typhus infection is highly focal This makes it difficult to define a target population for the purpose of making inferences. We will define the target population in terms of the village level sero-prevalence. The aim is to correlate the incidence of scrub typhus with the sero-prevalence at village level. This will allow using the results of the study to predict the expected incidence and burden of scrub typhus in other settings with a known sero-prevalence, and eventually estimate the global burden of scrub typhus (not part of the study but a potential extension of the work). The target population for the study is therefore "villages in which the IgG sero-prevalence is at least 15%".

ELIGIBILITY:
Inclusion Criteria:

* General population cohort: residing in study villages
* serological cohort: aged 10 years or older
* Hospital cohort: all ages

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General population cohort: all residents in scrub typhus endemic villages Serological cohort: random sample of 4000 individuals older than 10 years present at the time of the initial baseline survey visit
  hospital case cohort: cases of all ages attending study clinics for undifferentiated fever of at least 5 days duration
Sampling Method: Non-Probability Sample
Enrollment: 32566 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of scrub typhus | 2 years
  clinically apparent infection
Incidence of spotted fever | 2 years
  clinically apparent infection
Incidence of murine typhus | 2 years
  clinically apparent infection

SECONDARY OUTCOMES:
Incidence of serological infection (scrub typhus) | 2 years
  measured using paired samples from sero-cohort
Incidence of serological infection (spotted fever) | 2 years
  measured using paired samples from sero-cohort
Incidence of serological infection (murine typhus) | 2 years
  measured using paired samples from sero-cohort
Incidence of complicated infection (scrub typhus) | 2 years
  based on pre-defined complications: ARDS, shock, CNS, renal failure, myocarditis
Incidence of complicated infection (spotted fever) | 2 years
  based on pre-defined complications: ARDS, shock, CNS, renal failure, myocarditis
Incidence of complicated infection (murine typhus) | 2 years
  based on pre-defined complications: ARDS, shock, CNS, renal failure, myocarditis

CONTACTS AND LOCATIONS:
Overall Officials: Wolf-Peter Schmidt, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Daniel Chandramohan, PhD, Study Chair — London School of Hygiene and Tropical Medicine
Locations (1):
- Christian Medical College, Vellore, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Yes
de-identified case data will be made available at LSHTMs data repository
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: from 12/2022 indefinitely
Access Criteria: on request
URL: https://datacompass.lshtm.ac.uk

REFERENCES:
- [Derived] Devamani C, Alexander N, Chandramohan D, Stenos J, Cameron M, Abhilash KPP, Mangtani P, Blacksell S, Vu HTT, Rose W, Schmidt WP. Incidence of Scrub Typhus in Rural South India. N Engl J Med. 2025 Mar 13;392(11):1089-1099. doi: 10.1056/NEJMoa2408645. PMID 40073309

DOCUMENTS (2):
  • Study Protocol (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT04506944/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT04506944/SAP_001.pdf